CLINICAL TRIAL: NCT02652494
Title: Observational Study of Apremilast Use and Effectiveness Over a One Year Treatment Period in Patients With Psoriasis in The Netherlands
Brief Title: Observational Study of Apremilast in Patients With Psoriasis in The Netherlands
Acronym: APRIL
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-10004-PSOR-014
Record Dates: First submitted 2016-01-08; First posted 2016-01-12 (Estimated); Last update posted 2024-05-13 (Actual); Status verified 2020-07

CONDITIONS: Psoriasis
Keywords: Psoriasis; Observational; Apremilast; APRIL; Non-Interventional; The Netherlands
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients receiving Apremilast per daily clinical practice: Dutch patients receiving Apremilast according to daily clinical practice

SUMMARY:
This is a multicenter, prospective, non-interventional, observational single arm study.

Two-hundred patients will be recruited in the Netherlands over a one year period. In all cases, the decision to treat the patient with apremilast will be made prior to the decision to enter the subject into this study. Treatment will be according to routine clinical practice and based on recommendations as per the SPC of apremilast (Otezla®). Recruitment will continue until 200 patients have entered the study. Each patient will be followed for 12 months.

DETAILED DESCRIPTION:
Baseline Demographics, disease characteristics and medication history prior to start of treatment with apremilast will be collected. Patients will be asked to complete baseline DLQI, SF36, EQ5D, TSQM,WPAI and PBI questionnaires. Photographs of the finger nails will be taken.

Follow-up visits Follow-up assessments will take place at the regularly scheduled outpatient visits at 6 and 12 months (+/- 1 month) after initiation of apremilast.

* Skin-specific disease measures (Psoriasis Activity and Severity Index (PASI), (static) Physician Global Assessment (sPGA), Body Surface Area (BSA))
* Patients will be asked to complete the following questionnaires:
* DLQI
* TSQM
* EQ5D
* SF36- Itch Visual Analog Scale (VAS)
* WPAI Work Productivity and Activity Index
* Patient Benefit Index PBI

End of treatment Upon discontinuation of treatment with apremilast, the date, the dose and reason for discontinuation will be documented.

AE monitoring All patients will be monitored for adverse events throughout the study.

From the time of the patient signing informed consent until treatment with apremilast is permanently abrogated, all non-serious adverse events that are considered related to apremilast and all Serious Adverse Events (SAEs) regardless of causality will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age who understand and voluntarily sign an informed consent form.
* Patients starting treatment for psoriasis with apremilast in clinical practice.

Exclusion Criteria:

* Refusal to participate in the study.
* Women who are pregnant or breast-feeding.
* Hypersensitivity to the active substance or to any of the excipients.
* Prior exposure to apremilast
* Psoriatic arthritis treated by a rheumatologist in the previous year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two hundred adult patients treated with apremilast for psoriasis in clinical practice. In all cases, the decision to treat the patient with apremilast will be made prior to the decision to enter the subject into the study.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with Dermatology Life Quality Index (DLQI) ≤ 5 points | Up to approximately 12 months
  The Dermatology Life Quality Index or DLQI is a dermatology-specific Quality of Life instrument. It is a simple 10-question validated questionnaire that has been used in over 40 different skin conditions.
Percentage of patients with Dermatology Life Quality Index (DLQI) improvement in DLQI ≥ 5 points | Up to approximately 12 months
  The Dermatology Life Quality Index or DLQI is a dermatology-specific Quality of Life instrument. It is a simple 10-question validated questionnaire that has been used in over 40 different skin conditions.

SECONDARY OUTCOMES:
Changes in treatment satisfaction questionnaire for medication (TSQM) at 6 and 12 months treatment | Up to approximately 12 months
  The TSQM questionnaire is a general measure of treatment satisfaction across medication types and patient conditions.
Changes in generic quality of life at 6 and 12 months treatment Short Form 36 (SF-36v2) health survey | Up to approximately 12 months
  The SF-36v2® Health Survey measures functional health and well-being from the patient's point of view. It can be used across age (18 and older), disease, and treatment group.
Changes in generic quality of life at 6 and 12 months treatment using EuroQol-5 dimensions (EQ-5D) | Up to approximately 12 months
  EQ-5D is a standardized instrument for use as a measure of health outcome in a wide range of health conditions and treatment
Change in itch at 6 and 12 months treatment using the itch Visual Analog Scale (VAS) | Up to approximately 12 months
  Itch VAS is a simple assessment of the itch severity using a visual analogue scale
Changes in psoriasis area and severity index (PASI) at 6 and 12 months treatment | Up to approximately 2 months
  PASI score is a tool used to measure the severity and extent of psoriasis (Psoriasis Area and Severity Index).
Changes in body surface area (BSA)at 6 and 12 months treatment | Up to approximately 12 months
  BSA (Body Surface Area): severity is defined by how much of the body surface area is affected.
Changes in static physician global assessment (sPGA) at 6 and 12 months treatment | Up to approximately 12 months
  sPGA: assessment by physician to classify disease activity in a consistent manner
Baseline characteristics of patients initiating apremilast treatment | Up to approximately 1 month
  Characteristics at baseline of patient initiating apremilast treatment
Reasons for discontinuation of apremilast | Up to approximately 12 months
  Rate and reasons for discontinuation of apremilast within 12 months of start

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (12):
- Netherlands (12):
  - Zorggroep Twente, Hengelo, Gelderland
  - Radboud UMC, Nijmegen, Gelderland
  - Zuyderland MC, Sittard, Limburg
  - Bravis Ziekenhuis, Bergen op Zoom, North Brabant
  - Amphia, Breda, North Brabant
  - TweeSteden Ziekenhuis, Tilburg, North Brabant
  - Maxima MC, Veldhoven, North Brabant
  - Centrum Oosterwal, Alkmaar, North Holland
  - Spaarne Gasthuis, Hoofddorp, North Holland
  - Antonius Ziekenhuis Sneek, Sneek, Provincie Friesland
  - Maasstad Ziekenhuis, Rotterdam, South Holland
  - Meander MC, Amsersfoort, Utrecht

REFERENCES:
- [Background] van den Reek JMPA, van der Leest RJT, Thomas SE, Prevoo R, Plantenga ME, de Jong EMGJ. Improved Quality of Life in Patients with Psoriasis Receiving Apremilast: Real-World Data from the Netherlands. Adv Ther. 2024 Apr;41(4):1594-1605. doi: 10.1007/s12325-023-02759-9. Epub 2024 Feb 24. PMID 38402373
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Expanded Access for CC-10004 — https://clinicaltrials.gov/ct2/show/NCT02652494?term=CC-10004-PSOR-014&rank=1